CLINICAL TRIAL: NCT05567861
Title: Observational Study on the Effect of Virtual Reality on the Pain Intensity of Patients Suffering From Fibromyalgia
Brief Title: Virtual Reality for Fibromyalgia
Acronym: VR_Fibro
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 22-20
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Virtual Reality; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fibromyalgia is a frequent chronic pain syndrome almost often affecting women and associating diffuse chronic musculoskeletal pain (for more than 3 months), fatigue and sleep disturbances. Other varied functional symptoms are associated with it, in particular cognitive disorders and a feeling of unrested awakening.

Technological advances in virtual reality have led to recognition by the medical community as a way to improve pain and quality of life for patients.

There is a growing body of evidence supporting the use of virtual reality as an adjunct therapy to reduce acute pain in patients during medical procedures in hospital settings. There may also be a role for virtual reality in patients with chronic pain.

DETAILED DESCRIPTION:
Current treatments for fibromyalgia (FM) include pharmaceutical pain medications as well as psychological programs with components of cognitive therapy, and activity management. However, pain medications are not fully effective, can be addictive, and can cause hyperalgesia. Non-pharmacological treatments for chronic pain may be associated with limiting side effects, technology-based interventions using virtual reality (VR) may be a promising alternative treatment option.

There is evidence which shows that VR can be an effective treatment for pain reduction. However, most studies which utilize VR as a method of pain reduction focus on acute pain and studies looking at VR for chronic pain are scarce.

Investigator will analyze the pain reduction and impact on behavioral mechanisms and cognition with repetitive active VR on Fibromyalgia

ELIGIBILITY:
Inclusion Criteria :

* Patients able to understand and sign the informed consent form for the study
* Adults aged 18 to 65 years
* Followed in algology for fibromyalgia pain > 6 months
* With mean pain intensity ≥ 4

Exclusion Criteria :

* History of epilepsy or hypersensitivity to flashing light to limit the risk of virtual reality-induced seizures
* Previous use of VR for pain (possible bias)
* Refusal to participate
* Therapeutic modifications for pain management related to fibromyalgia during the first month of participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with fibromyalgia pain > 6 months
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Patient pain | month 1
  Numerical Rating Scale, 0 to 10, 0 = no pain, 10 = maximal pain

SECONDARY OUTCOMES:
Patient pain | week 2, month 2
  Numerical Rating Scale, 0 to 10, 0 = no pain, 10 = maximal pain
Activity | month 1, month 2
  pain self-efficacy questionnaire, 0 to 60, 0 = not at all confident, 60 = completely confident
Mood | month 1, month 2
  Hospital Anxiety and Depression scale, 0 to 42, 7 or less = no symptom, 8 to 10 = doubt on symptom, 11 and more = undeniable symptom
Pain associated cognition | month 1, month 2
  Catastrophizing scale, 0 to 52, higher score indicates higher level of catastrophizing, a total score above 30 indicates clinically relevant level of catastrophizing

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco